CLINICAL TRIAL: NCT06975293
Title: Open-label, Non-randomized, Multi-cohort, Phase 1b/2 Trial Investigating the Safety, Tolerability, and Antitumor Activity of STC-15 (a METTL3 Inhibitor) as a Part of Combination Therapy With Toripalimab in Participants With Selected Advanced Cancers
Brief Title: STC-15 as a Part of Combination Therapy With Toripalimab in Selected Advanced Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: STORM Therapeutics LTD (Industry)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STC-15-24202
Record Dates: First submitted 2025-04-14; First posted 2025-05-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Non-small Cell Lung Cancer; Metastatic Melanoma; Metastatic Endometrial Cancer; Metastatic Head-and-neck Squamous-cell Carcinoma; Solid Tumor
Keywords: STC-15; Toripalimab; PD1; Checkpoint Combination
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose escalation (Experimental): Phase 1b 3+3 trial design of dose escalation of STC-15 in combination with toripalimab
  Interventions: Combination Product: STC-15 in combination with toripalimab
- Dose expansion NSCLC (Experimental): STC-15 in combination with toripalimab (anti-PD-1) in locally advanced and unresectable or metastatic NSCLC
  Interventions: Combination Product: STC-15 in combination with toripalimab
- Dose expansion melanoma (Experimental): STC-15 in combination with toripalimab in locally advanced unresectable or metastatic melanoma
  Interventions: Combination Product: STC-15 in combination with toripalimab
- Dose expansion endometrial cancers (Experimental): STC-15 in combination with toripalimab in locally advanced unresectable or metastatic endometrial cancers
  Interventions: Combination Product: STC-15 in combination with toripalimab
- Dose expansion HNSCC (Experimental): STC-15 in combination with toripalimab in locally advanced or metastatic HNSCC
  Interventions: Combination Product: STC-15 in combination with toripalimab

INTERVENTIONS:
Combination Product: STC-15 in combination with toripalimab — STC-15 in combination with toripalimab in 21-day cycles

SUMMARY:
This early phase oncology trial will be conducted at various study centers to investigate the safety, tolerability, and antitumor activity of STC-15 (a METTL3 inhibitor) in combination with toripalimab (anti- programmed cell death 1 [PD-1]) in four different locally advanced unresectable or metastatic tumors such as indications: (1) in combination with toripalimab (anti- programmed cell death 1 [PD-1]) in locally advanced and unresectable or metastatic non-small cell lung cancer (NSCLC), (2) in combination with toripalimab in locally advanced unresectable or metastatic melanoma, (3) in combination with toripalimab in locally advanced unresectable or metastatic endometrial cancers, and (4) in combination with toripalimab in locally advanced or metastatic head and neck squamous cell carcinoma (HNSCC).

This study comprises of 2 parts: a combination dose escalation part (Phase 1b) followed by an assessment of the combination treatment's antitumor activity (Phase 2). This study will be conducted in adult participants with advanced malignancies to characterize the safety, tolerability, PK, and clinical activity of STC-15 in combination with toripalimab.

ELIGIBILITY:
Key Inclusion Criteria:

* Estimated life expectancy ≥ 3 months.
* ECOG performance status 0 or 1.
* Measurable disease according to RECIST v1.1 as assessed by the local site investigator/radiology.
* Documented radiologic assessment of progression on the prior therapy before study entry.
* Have the ability to swallow, retain, and absorb oral medication.

Inclusion Criteria (Expansion):

* NSCLC (when applicable): Participants with AGAs (actionable genetic alterations) must have received targeted therapy unless contraindicated. Participants must not have received more than three previous lines of systemic treatment for unresectable locally advanced or metastatic disease. This must include at least a prior anti-PD-1/L1 alone or in combination with chemotherapy. Participants must have disease progression on prior anti-PD-1/L1.
* HNSCC (when applicable): Participants must have progressed on following prior lines: 2L or 3L recurrent/metastatic disease; regardless of PD-L1 score. Participants must not have received more than three previous lines of systemic treatment for unresectable locally advanced or metastatic disease. This must include at least a prior anti-PD-1/L1 alone or in combination with chemotherapy.
* Endometrial (when applicable): Participants must not have received more than three previous lines of systemic treatment for unresectable locally advanced or metastatic disease. This must include at least a prior anti-PD-1/L1 alone or in combination with chemotherapy. Participants must have disease progression on prior anti-PD-1/L1
* Melanoma (when applicable): Participants must not have received more than three previous lines of systemic treatment for unresectable locally advanced or metastatic disease. This must include at least a prior anti-PD-1/L1 alone or in combination with chemotherapy. Participants must have disease progression on prior anti-PD-1/L1.

Key Exclusion Criteria:

* Pregnant and lactating women.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks prior to first IMP administration.
* Participants who have not recovered from all AEs due to previous therapies to Grade ≤ 1 or baseline, according to NCI-CTCAE v5.0. Exceptions include: alopecia, Grade ≤ 2 neuropathy, and endocrine-related AEs Grade ≤ 2 who are stable on treatment or hormone replacement.
* Major surgery less than 4 weeks prior to the first IMP administration or participants who have not recovered from the side effects of the surgery.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or the presence of ongoing pneumonitis/interstitial lung disease).
* Clinically significant cardiovascular disease or condition.
* Known active CNS metastases and/or leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of STC-15 in combination with toripalimab | 6 months
  Incidence of adverse events graded according to CTCAE v5.0

SECONDARY OUTCOMES:
Anti-tumor activity | 6 months
  To evaluate the antitumor activity of STC-15 in combination with toripalimab as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST) criteria
Maximum observed plasma concentration of STC-15 (Cmax) | 22 days
Recommended Phase 2 Dose | 6 months
  Identification of a tolerable and safe dose for expansion cohorts based on dose limiting toxicities
Calculated time to reach maximum observed plasma concentration (Tmax) | 22 days
Calculated area under the plasma concentration-time curve of STC-15 (AUC0-t) | 22 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwell Health Cancer Institute, Lake Success, New York
  - The START Center, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided